CLINICAL TRIAL: NCT04430465
Title: Effects of Wholegrains on Children's Health (KORN)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Chalmers University of Technology (Other)
Responsible Party: Principal Investigator, Camilla Trab Damsgaard, Associate Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: D225
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-01

CONDITIONS: Cardiometabolic Health; Gastro-intestinal Wellbeing; Cognitive Function; Overweight
Keywords: Children; Wholegrain; Cardiovascular risk markers; Overweight; Adolescents
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The intervention and data collection will be conducted unmasked. The data set will be masked before data analysis by staff not involved in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High wholegrain then low wholegrain (Experimental): Starting with high wholegrain intervention followed by low wholegrain intervention
  Interventions: Dietary Supplement: Grain products high in wholegrains from oat and rye; Dietary Supplement: Grain products low in wholegrains
- Low wholegrain then high wholegrain (Experimental): Starting with low wholegrain intervention followed by high wholegrain intervention
  Interventions: Dietary Supplement: Grain products high in wholegrains from oat and rye; Dietary Supplement: Grain products low in wholegrains

INTERVENTIONS:
Dietary Supplement: Grain products high in wholegrains from oat and rye — A selection of grainproducts high in wholegrain from oat and rye, including cereals, bread, rolls, and pasta is replacing habitual grain products
  Other Names: Wholegrain
Dietary Supplement: Grain products low in wholegrains — A selection of grainproducts low in wholegrain, including cereals, bread, rolls, and pasta is replacing habitual grain products
  Other Names: Refined grain

SUMMARY:
KORN investigates the effects of wholegrain oat and rye intake on health and cognitive wellbeing in children with overweight.

DETAILED DESCRIPTION:
The purpose of KORN is to investigate the effects of wholegrain oat and rye intake on cardiometabolic health in slightly overweight 8-13-year-old children. Moreover, KORN aims to investigate effects on body weight and body composition, inflammatory markers, gastrointestinal wellbeing and cognitive function and explore the potential underlying mechanisms through assessment of changes in the children's gut microbiota as well as potential genotype-dependent and sex-specific effects.

The study has a randomized controlled cross-over design. In two 8-week dietary periods the children will receive grain products (cereals, breads, pasta etc) with either high or low content of wholegrain from oat and rye in random order. Measurements and biological sampling will be performed at 0, 8 and 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls 8-13 years of age
* Be overweight i.e. have a parent-reported BMI of at least +1 standard deviation above the median according to the age and sex-standardized Danish growth curves
* Be healthy
* Like grain products and eat them daily
* Speak Danish in order to understand the study procedures
* At least one parent must read and speak Danish, in order to be properly informed about the study procedures
* Parents must have freezer capacity for 2 weeks bread provision

Exclusion Criteria:

* Allergy or intolerance to the study foods, including gluten
* Use of dietary fiber supplements (e.g. HUSK) or probiotic supplements
* Dieting or on a special diet
* Serious chronic illnesses and diseases that may interfere with study outcomes
* Use of medication that may affect study outcomes, including use of antibiotics the last month
* Concomitant participation in other studies involving dietary supplements, drugs or blood sampling
* Living in a household with another participating child

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-05-04 (Actual)

PRIMARY OUTCOMES:
Low density lipoprotein cholesterol | 16 weeks
  by fasting blood sample
Insulin | 16 weeks
  by fasting blood sample

SECONDARY OUTCOMES:
Height | 16 weeks
  by stadiometer
Weight | 16 weeks
  by digital scale
Body Mass Index z-score | 16 weeks
  by height and weight measurements
Waist circumference | 16 weeks
  by measuring tape
Fat mass index | 16 weeks
  by Dual-energy X-ray Absorptiometry
Fat free mass index | 16 weeks
  by Dual-energy X-ray Absorptiometry
Systolic blood pressure | 16 weeks
  by digital device
Diastolic blood pressure | 16 weeks
  by digital device
Heart rate | 16 weeks
  by digital device
Glucose | 16 weeks
  by fasting blood sample
Glycosylated hemoglobin (HbA1c) | 16 weeks
  by fasting blood sample
Triacylglycerol | 16 weeks
  by fasting blood sample
High density lipoprotein cholesterol | 16 weeks
  by fasting blood sample
Total cholesterol | 16 weeks
  by fasting blood sample
High sensitivity C-reactive protein | 16 weeks
  by fasting blood sample
Attention | 16 weeks
  assessed by d2 test of attention
Inhibition | 16 weeks
  assessed by Stroop color and word test
Processing speed | 16 weeks
  assessed by d2 test of attention and Stroop color and word test
Working memory | 16 weeks
  assessed by Kim's game
Socio-emotional skills | 16 weeks
  assessed by parent reported Strengths and Difficulties Questionnaire
Stool consistency | 16 weeks
  assessed by the Bristol stool scale
Gastrointestinal wellbeing | 16 weeks
  assessed by questionnaire
Prevalence of overweight | 16 weeks
  By the International Obesity Task Force criteria

OTHER OUTCOMES:
Dietary intake | 16 weeks
  assessed by 4-day dietary record
Physical activity | 16 weeks
  assessed by questionnaire
Sociodemographic characteristics | at baseline
  assessed by questionnaire
Pubertal development stage | at baseline
  assessed by the Tanner scales
General satisfaction | 16 weeks
  assessed by questionnaire
Liking of study products | 16 weeks
  assessed by questionnaire
Alkylresorcinols (compliance) | 16 weeks
  by fasting blood sample
Android fat mass index | 16 weeks
  by Dual-energy X-ray Absorptiometry
Gynoid fat mass index | 16 weeks
  by Dual-energy X-ray Absorptiometry
Android:gynoid fat mass ratio | 16 weeks
  by Dual-energy X-ray Absorptiometry
Immune cell count | 16 weeks
  by fasting blood sample
Interleukin 6 (IL-6) | 16 weeks
  by fasting blood sample
Interleukin 1β (IL-1β) | 16 weeks
  by fasting blood sample
Tumor necrosis factor alpha (TNFα) | 16 weeks
  by fasting blood sample
Bone Mineral Density | 16 weeks
  by Dual-energy X-ray Absorptiometry
Bone Mineral Content | 16 weeks
  by Dual-energy X-ray Absorptiometry
Bone area | 16 weeks
  by Dual-energy X-ray Absorptiometry
Gut microbiome composition determined by high throughput sequencing and qPCR | 16 weeks
  by fecal sample
Short chain fatty acids | 16 weeks
  by fasting blood sample
Short chain fatty acids | 16 weeks
  by fecal sample
Bile acids | 16 weeks
  by fasting blood sample
Bile acids | 16 weeks
  by fecal sample
Fatty acid composition | 16 weeks
  by fasting blood sample
C-peptide | 16 weeks
  by fasting blood sample
Epigenetics | 16 weeks
  by fasting blood sample
Metabolomics | 16 weeks
  by fasting blood sample
Metabolomics | 16 weeks
  by fecal sample
Proteomics | 16 weeks
  by fasting blood sample
Proteomics | 16 weeks
  by fecal sample
Genotypes | 16 weeks
  by fasting blood sample
Adiponectin | 16 weeks
  by fasting blood sample
Leptin | 16 weeks
  by fasting blood sample
Appetite hormones | 16 weeks
  by fasting blood sample
Testosterone | 16 weeks
  by fasting blood sample
Estrogen | 16 weeks
  by fasting blood sample
Gonadotropins | 16 weeks
  by fasting blood sample

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nutrition, Exercise and Sports, University of Copenhagen, Frederiksberg, Denmark

REFERENCES:
- [Derived] Madsen MTB, Landberg R, Nielsen DS, Zhang Y, Anneberg OMR, Lauritzen L, Damsgaard CT. Effects of Wholegrain Compared to Refined Grain Intake on Cardiometabolic Risk Markers, Gut Microbiota, and Gastrointestinal Symptoms in Children: A Randomized Crossover Trial. Am J Clin Nutr. 2024 Jan;119(1):18-28. doi: 10.1016/j.ajcnut.2023.10.025. Epub 2023 Oct 28. PMID 37898434